CLINICAL TRIAL: NCT06033417
Title: The Effect of an 8-week Walking Intervention on Blood Pressure in Older Adults With Respiratory Impairment: A Pilot Study.
Brief Title: Walking and Blood Pressure in Older Adults With Respiratory Impairment.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Iowa State University (Other)
Responsible Party: Principal Investigator, Duck-chul Lee, Professor, Kinesiology, Iowa State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-200-00
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Respiratory Impairment; Elevated Blood Pressure; Physical Inactivity
Keywords: Physical activity; Step counts; Lung function; Blood pressure; Older adults; Walking
MeSH Terms: conditions — Respiratory Insufficiency; Hypertension; Sedentary Behavior; Motor Activity | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Increased lifestyle walking (intervention) (Experimental): Intentional increase in daily steps: 3,000 extra steps/day, 5-days a week, 8-weeks total.
  Interventions: Other: Increased lifestyle walking (intervention)
- Health education only (control) (Other): Health education and no intentional increase in baseline daily steps (but with the option to receive the intervention upon conclusion of the initial 8-weeks).
  Interventions: Other: Health education only (control)

INTERVENTIONS:
Other: Increased lifestyle walking (intervention) — Participants will increase their baseline steps by a minimum of 3,000 extra steps/day, 5-days/week, for 8-weeks. Baseline steps will be assessed using a pedometer over a 7-day period before the intervention, after which a new (higher) daily step target will be assigned. The intervention will take place in the free-living setting, with participants reaching their step goals by engaging in more activities of daily living or via purposeful physical activity. Participants will wear a pedometer throughout the 8-week period to keep track of their steps, and adherence to the protocol will be determined by collecting the stored step data directly from each participant's pedometer on a weekly basis. Participants will be supported in their efforts to meet their daily step targets by engaging in once-weekly walking groups (30-mins/session) led by research staff. They will also receive 20-minute phone calls once every two weeks to set goals and create action plans for reaching their step targets.
  Arms: Increased lifestyle walking (intervention)
Other: Health education only (control) — Those randomized to the delayed participation group will be instructed to maintain their 'normal' lifestyle activities, thereby avoiding any significant increase in daily step counts beyond their 'baseline' values. Participants will wear a pedometer throughout the 8-week period to keep track of their steps, and adherence to the protocol will be determined by collecting the stored step data directly from each participant's pedometer on a weekly basis. Participants in this group will attend once-weekly group health education sessions (30-minutes/session), in addition to 5-minute, 'touch base' phone calls once every 2-weeks, but these phone calls will not involve goal-setting or action planning. After completing the initial 8-week period, these individuals can then opt to undertake the 'increased lifestyle walking' intervention of 3,000 extra steps/day over 5-days for 8-weeks if desired.
  Arms: Health education only (control)

SUMMARY:
The purpose of this study is to evaluate the effect of an 8-week walking program on blood pressure in inactive older adults with respiratory impairment, a condition where lung function is sub-optimal for a person's age. Older adults with respiratory impairment have greater risks of death by cardiovascular disease (CVD) compared to those without respiratory impairment, and this may be partly driven by higher resting blood pressure. One way to lower blood pressure is to increase the number of daily steps achieved throughout the course of everyday life ('lifestyle steps'), and previous research shows that an additional 3,000 lifestyle steps/day is effective for achieving this. However, whether an increase in daily lifestyle steps is effective for reducing blood pressure in senior-community dwelling older adults with respiratory impairment is unknown. Understanding how increasing daily steps impacts blood pressure in this understudied population is important for informing future strategies for tackling cardiovascular disease risk in those with lung dysfunction.

DETAILED DESCRIPTION:
Older adults are particularly susceptible to respiratory impairment (a condition of lung dysfunction) due in part to longer lifetime exposures to air pollutants, tobacco smoke, and physical inactivity. Older adults with respiratory impairment have greater long-term risks of death by cardiovascular disease (CVD) when compared to individuals without respiratory impairment. Impaired lung function tends to run parallel with high blood pressure, and high blood pressure is a determinant of CVD mortality in this population. One approach to lowering blood pressure across the lifespan is by increasing physical activity (PA) behavior. Walking is the most commonly practiced modality of PA in older adulthood, and previous studies show that accumulating an additional 3,000 steps/day over 5-days a week through activities of daily living (i.e., 'lifestyle stepping') reduces blood pressure in inactive older adults free from respiratory impairment. This step-based PA prescription roughly equates to 150-minutes of moderate-intensity aerobic PA/week for most inactive older adults, and therefore satisfies the minimum aerobic PA recommendations for substantial health benefits. However, the impact of such an intervention on blood pressure in older adults with respiratory impairment is unclear. The 'Physical Activity Guidelines for Americans: Midcourse Report' (2023) indicates that senior centers are key settings for successful PA interventions. Senior-living communities are traditionally well-designed and well-resourced to support PA (e.g., safe outdoor walking spaces; access to indoor exercise facilities; social support, etc.), making them highly suitable locations for lifestyle walking. Additionally, the prescription of PA using lifestyle step counts rather than time-based prescriptions is intuitive and arguably easier to integrate into activities of daily living. However, no study has yet evaluated the effect of increasing daily lifestyle step counts on blood pressure in older adults with respiratory impairment. Addressing this gap in knowledge will provide support for the utility of lifestyle walking as a therapeutic approach to CVD risk management in older adults with lung dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 65 years and above.
* Elevated systolic blood pressure (120mmHg - 159 mmHg), and/or individuals taking medications for high blood pressure with a systolic pressure less than or equal to 159mmHg.
* Respiratory impairment as assessed by abnormal spirometry (a lung function test). Abnormal spirometric phenotypes include obstructive pattern, restrictive pattern, mixed obstructive/restrictive, and preserved ratio impaired spirometry (PRISm).
* Non-smoker (defined as being tobacco-free for at least the previous 12-months).
* Body mass index (BMI) <42kg/m2.
* Physically inactive (determined by a 7-day day assessment of step counts using a pedometer, and defined as having an average daily step count <7,000).
* Willingness to increase daily steps.

Exclusion Criteria:

* History of stroke, heart attack, or cancer diagnosis in the last 6-months.
* Admission to hospital for a respiratory-related illness (e.g., COPD exacerbation, pneumonia, lung injury, etc.) within the last 3 months.
* The use of supplemental oxygen.
* Neurological conditions such as Alzheimer's or Parkinson's disease.
* Significant mobility limitation (e.g., severe arthritis) that would hinder the ability to increase daily steps.
* The use of a cane or walker.
* Participants engaged in another walking study or structured walking program.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Change in systolic blood pressure | 0-weeks, 8-weeks
  Pre- and post-intervention brachial blood pressure (upper left arm) will be assessed after 10-minutes of quiet rest in the supine position using the SphygmoCor device (AtCor Medical, Itasca, IL, USA), an automated blood pressure monitor. The participant will be free of constrictive clothing, their legs will be uncrossed, and their back will be supported by a cushioned surface (i.e., bed) beneath them. A minimum of 3 blood pressure measurements will be taken at intervals of at least 2 minutes.

SECONDARY OUTCOMES:
Feasibility of conducting the study | 8-weeks
  The secondary purpose of this pilot study is to explore two (2) facets of feasibility: adherence and attrition, with the study considered to be feasible if 'high adherence' and 'low attrition' are observed. High adherence is defined as all participants meeting their daily step goals 80% of the time (i.e., 32 days out of a possible 40 days). Low attrition is defined as 80% or more participants attending both pre- and post-intervention assessments.

OTHER OUTCOMES:
Change in arterial stiffness | 0-weeks, 8-weeks
  Pre- and post-intervention arterial stiffness will be estimated through the assessment of carotid-femoral pulse wave velocity using the SphygmoCor device (AtCor Medical, Itasca, IL, USA) immediately following the resting blood pressure assessment. The participant will lie down and a blood pressure cuff will be placed around the upper leg and a pressure sensor will be applied to the carotid artery to obtain femoral and carotid pulse waves. The distance between the femoral and carotid pulses will be measured with a tape measure and the pulse transit time between the two locations will be calculated by the SphygmoCor device (AtCor Medical, Itasca, IL, USA).
Change in lung function | 0-weeks, 8-weeks
  Pre- and post-intervention lung function will be assessed by spirometry using a handheld spirometer (EasyOne Air, NDD Medical Technologies, Andover, MA), specifically performing the Forced Vital Capacity (FVC) maneuver. The participant begins by inhaling air to maximum lung volume without the device in their mouth, and then forcefully exhaling through the device until the lungs are completely emptied. A minimum of 3 and a maximum of 8 FVC maneuvers will be will be performed following the American Thoracic Society guidelines, and the device will use inbuilt algorithms to measure the forced expiratory time. The primary indices of lung function will include the Forced Vital Capacity (FVC), the Forced Expiratory Volume in 1-second (FEV1), and the ratio between the two (FEV1/FVC).
Change in SPPB performance | 0-weeks, 8-weeks
  Pre- and post-intervention assessment of lower extremity functioning consists of a usual-paced walking test (i.e., normal gait speed) over a flat 4m course; a series of two-footed balance poses each lasting 10 seconds: feet side-by-side, feet partially staggered [semi-tandem], and feet in the heel-to-toe position [fully tandem]; and five unaided chair stands completed as quickly as possible.
Change in functional capacity | 0-weeks, 8-weeks
  Pre- and post-intervention functional capacity will be evaluated using the fast 400m walk test, a validated measure of walking ability and endurance designed specifically for older adults. Participants will walk at a fast pace around two cones set 20m apart in a long hallway on level ground for 10 full laps (i.e., 400m), and the time taken to complete the test (mins:secs) will be recorded (faster times equate to better functional capacity). Participants will be provided with verbal encouragement throughout to test to maximize the effort exerted.
Change in exertional dyspnea (breathlessness) | 0-weeks, 8-weeks
  Pre- and post-intervention exertional dyspnea (the perception of breathlessness experienced during exercise) will be assessed using a validated 10-level severity scale (modified Borg index) where 0 = no shortness of breath and 10 = maximum shortness of breath. The Borg index will be administered immediately following completion of the functional capacity test (i.e., fast 400m walk).
Change in sleep quality | 0-weeks, 8-weeks
  Pre- and post-intervention sleep quality will be evaluated using the validated Pittsburgh Sleep Quality Index (PSQI).
Change in quality of life | 0-weeks, 8-weeks
  Pre- and post-intervention quality of life will be evaluated using the validated 36-item short form survey (SF-36).
Change in respiratory symptoms | 0-weeks, 8-weeks
  Pre- and post-intervention respiratory symptoms will be evaluated using the validated St. George's Respiratory Questionnaire (SGRQ).
Change in fatigability | 0-weeks, 8-weeks
  Pre- and post-intervention physical and mental fatigability will be evaluated using the validated Pittsburgh Fatigability Scale. This is a 10-item questionnaire that evaluates self-reported whole-body physical and mental tiredness anchored to activities of fixed intensity and duration in adults age ≥60 years. Each item in the scale ranges from 0 to 5, where 0 represents "no fatigue whatsoever" and 5 represents "extreme fatigue." The scores from each item are then summed to give a total score between 0 and 50. A higher score reflects greater fatigability.
Change in cognitive performance | 0-weeks, 8-weeks
  Pre- and post intervention cognitive performance will be evaluated using the validated modified mini-mental state examination (3MS).
Change in waist circumference | 0-weeks, 8-weeks
  Pre- and post intervention waist circumference (measured in cm) will be evaluated using a digital measuring tape (Smart Tape Measure V001, Fitindex, Eastvale, CA).

CONTACTS AND LOCATIONS:
Overall Officials: Duck-chul Lee, PhD, Principal Investigator — Iowa State University
Locations (1):
- Iowa State University, Ames, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified, individual participant data may be shared with researchers outside of the institution upon submission of a pre-analysis plan and, if required by federal regulations, approval from the institutional review board (IRB).
Supporting Information: Study Protocol
Time Frame: Data will become available for sharing from January 2024 onward, and pre-analysis plans can be submitted indefinitely thereafter.
Access Criteria: There are no data-sharing agreements in place at this time. However, the study has IRB support to share data in a manner that maintains the confidentiality of participants, honors assurances made to participants during informed consent, and complies with data privacy regulations. Researchers wishing to affiliate with the project must first pass a course on the Protection of Human Subjects, and data requests will be conveyed to the institutional review board (IRB) (if required). The IRB will determine the nature of the request and later provide recommendations. Approval will be based on a pre-submitted analysis plan from the researchers. Upon approval, an agreement between the PI and the researchers will be made, and de-identified data will be cut from the main dataset and distributed electronically. The researchers will agree to publish only the results of the analysis plan, and must seek further assent if significant deviations from this plan are made.